CLINICAL TRIAL: NCT00190476
Title: Randomized Controlled Trial Comparing Docetaxel-cisplatin Combination With Docetaxel Alone in Elderly Patients With Advanced Non-small-cell Lung Cancer(JCOG0207)
Brief Title: Elderly NSCLC/D vs DP (JCOG0207)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Japan Clinical Oncology Group (Other)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JCOG0207; C000000146
Record Dates: First submitted 2005-09-11; First posted 2005-09-19 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Non-small-cell Lung Cancer
Keywords: Elderly; advanced; non-small-cell lung cancer; cisplatin; docetaxel; weekly; combination; chemotherapy; randomized trial
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Weekly docetaxel alone
Drug: Weekly docetaxel + cisplatin combination

SUMMARY:
To evaluate the efficacy of docetaxel-cisplatin combination in comparison to docetaxel alone for elderly patients with advanced non-small-cell lung cancer.

DETAILED DESCRIPTION:
The Elderly Lung Cancer Vinorelbine Italian Study demonstrated the first evidence of the utility of chemotherapy in elderly patients with advanced non-small-cell lung cancer (NSCLC). In a large randomized trial, gemcitabine and vinorelbine failed to show any advantage over either agent alone. With the current evidence, single agent chemotherapy with a third-generation drug can be considered a recommended option for elderly patients with advanced NSCLC. A Japanese phase I/II study showed the activity (overall response rate 52%, median survival 12.4 months) and tolerability of weekly docetaxel/ cisplatin combination in patients older than age 75 years. There have been no randomized prospective trials dedicated to elderly NSCLC patients to evaluate tolerability and efficacy of platinum-based combination.

Comparison: Single-agent weekly docetaxel versus weekly regimen of docetaxel-cisplatin combination for elderly advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. histologically or cytologically proven non-small-cell lung cancer
2. stage IV, or stage III disease ineligible for definitive radiotherapy
3. 70 years or older
4. ECOG PS 0-1
5. Ineligible for standard platinum(bolus infusion)-containing combination chemotherapy
6. No prior chemotherapy(containing gefitinib) for non-small cell lung cancer or other neoplasms
7. No prior surgery within 4 weeks before enrollment
8. No prior radiotherapy for primary tumor
9. No prior radiotherapy for metastatic lesions within 2 weeks before enrollment
10. Adequate organ function
11. Signed informed consent

Exclusion Criteria:

1. Symptomatic brain metastasis
2. Active another neoplasms
3. Severe SVC syndrome
4. Massive pericardial, pleural effusion, or ascites
5. Bone metastasis emergent for palliative radiotherapy or surgery
6. Uncontrollable systemic hypertension
7. Heart failure, Unstable angina, Myocardial infarction within 6 months
8. Uncontrollable diabetes
9. Active infection
10. Interstitial pneumonia/ Pulmonary fibrosis
11. Hypersensitivity for polysorbate 80
12. Systemic administration of corticosteroids

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 230
Dates: Start 2003-04; Study Completion 2007-04

PRIMARY OUTCOMES:
overall survival

SECONDARY OUTCOMES:
Toxicity
Progression-free survival
Response rate
Symptom score

CONTACTS AND LOCATIONS:
Overall Officials: Akira Yokoyama, MD, PhD, Study Chair — Department of Internal Medicine, Niigata Cancer Center Hospital
Locations (29):
- Japan (29):
  - Aichi Cancer Center Hospital, Nagoya,Chikusa-ku,Kanokoden,1-1, Aichi-ken
  - Aichi Cancer Center,Aichi Hospital, Okazaki,Kake-machi,Kuriyado,18, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa,Kashiwanoha,6-5-1, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama,Horinouchi,13, Ehime
  - Kyushu University Hospital, Higashi-ku,Maidashi,3-1-1, Fukuoka
  - Gifu Municipal Hospital, Gifu,Kashima-cho,7-1, Gifu
  - Gunma Prefectural Cancer Center, Ota,Takabayashi-nishi-cho,617-1, Gunma
  - National Nishigunma Hospital, Shibukawa,Kanai,2854, Gunma
  - National Hospital Organization, Dohoku National Hospital, Asahikawa,Hanasaki,7-4048, Hokkaido
  - National Hospital Organization Hokkaido Cancer Center, Sapporo,Shiroishi-ku,Kikusui,4-2-3-54, Hokkaido
  - Hyogo Medical Center for Adults, Akashi,Kitaouji-cho,13-70, Hyōgo
  - Hyogo College of Medicine, Nishinomiya,Mukogawa-cho,1-1, Hyōgo
  - Ibaraki Kenritsu Chuo Hospital & Cancer Center, Nishi-ibarakigun,Tomobemachi,Koibuchi,6528, Ibaraki
  - Kanagawa Cancer Center, Yokohama,Asahi-ku,Nakao,1-1-2, Kanagawa
  - Yokohama Mucipical Citizen's Hospital, Yokohama,Hodogaya-ku,Okazawa-cho,56, Kanagawa
  - Kumamoto Regional Medical Center Hospital, Kumamoto,Honjo,5-16-10, Kumamoto
  - Niigata Cancer Center Hospital, Niigata,Kawagishi-cho, 2-15-3, Niigata
  - Osaka Prefectural Medical Center for Respiratory and Allergic Disease, Habikino,Habikino,3-7-1, Osaka
  - Osaka Medical Center for Cancer and Cardiovascular Diseases, Osaka,Higashinari-ku,Nakamichi,1-3-3, Osaka
  - Osaka City General Hospital, Osaka,Miyakojima-ku,Miyakojimahondori,2-13-22, Osaka
  - Kinki University School of Medicine, Osaka-Sayama,Ohno-higashi,377-2, Osaka
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Sakai,Nagasone,1180, Osaka
  - National Hospital Organization Toneyama National Hospital, Toyonaka,Toneyama,5-1-1, Osaka
  - Saitama Cancer Center, Kita-adachi,Ina,Komuro,818, Saitama
  - Sizuoka Cancer Center, Sunto-gun,Nagaizumi-cho,Shimonagakubo,1007, Shizuoka
  - Tochigi Cancer Center, Utsunomiya,Yohnan,4-9-13, Tochigi
  - National Cancer Center Hospital, Chuo-ku,Tsukiji,5-1-1, Tokyo
  - International Medical Center of Japan, Shinjuku-ku,Toyama,1-21-1, Tokyo
  - Yamagata Prefectural Central Hospital, Yamagata,Aoyagi,1800, Yamagata

REFERENCES:
- [Derived] Tsukada H, Yokoyama A, Goto K, Shinkai T, Harada M, Ando M, Shibata T, Ohe Y, Tamura T, Saijo N; Lung Cancer Study Group of the Japan Clinical Oncology Group (JCOG). Randomized controlled trial comparing docetaxel-cisplatin combination with weekly docetaxel alone in elderly patients with advanced non-small-cell lung cancer: Japan Clinical Oncology Group (JCOG) 0207dagger. Jpn J Clin Oncol. 2015 Jan;45(1):88-95. doi: 10.1093/jjco/hyu176. Epub 2014 Nov 6. PMID 25378648
- See also: Related Info — http://www.jcog.jp/